CLINICAL TRIAL: NCT02190019
Title: Transcranial Magnetic Stimulation for Apathy in Mild Cognitive Impairment:Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Prasad R. Padala, Associate Director for Clinical Programs, GRECC, Central Arkansas Veterans Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 391721
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Apathy; Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; apathy; executive function
MeSH Terms: conditions — Lethargy; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial magnetic stimulator (Active Comparator): Neurostar repetitive transcranial magnetic stimulator. The active procedure will stimulate at 120% motor threshold for 4 seconds at a frequency of 10 Hz, with an inter-train interval of 26 seconds for a total of 3,000 pulses. 10 treatment sessions are given over a two week period.
  Interventions: Device: Neurostar repetitive transcranial magnetic stimulator
- Sham coil treatment (Sham Comparator): Neurostar repetitive transcranial magnetic stimulator. 10 treatments identical in duration will be administered over a two week period.
  Interventions: Device: Neurostar repetitive transcranial magnetic stimulator

INTERVENTIONS:
Device: Neurostar repetitive transcranial magnetic stimulator — The active procedure will stimulate at 120% motor threshold for 4 seconds at a frequency of 10 Hz, with an inter-train interval of 26 seconds for a total of 3,000 pulses. 10 treatment sessions are given over a two week period.
  Other Names: rTMS

SUMMARY:
Mild cognitive impairment (MCI) is a precursor of dementia. Apathy, a profound loss of motivation, is a common behavioral problem in MCI. Presence of apathy may increase the chance of MCI patients converting to Alzheimer's Dementia. Repetitive Transcranial Magnetic Stimulation (rTMS), a non-invasive tool, has been recently approved for treatment of refractory depression. Since dysfunction in the frontal lobe of the brain is seen in patients with apathy, rTMS to the frontal lobe might be helpful in treating the same. Study hypotheses include that rTMS to the dorsolateral prefrontal cortex (DLPFC) will improve apathy and executive function better than sham treatment in those with MCI

DETAILED DESCRIPTION:
Objective: Mild cognitive impairment (MCI) is a precursor of dementia. Apathy, a profound loss of motivation, is a common behavioral problem in MCI. Presence of apathy may increase the chance of MCI patients converting to Alzheimer's Dementia. Repetitive Transcranial Magnetic Stimulation (rTMS), a non-invasive tool, has been recently approved for treatment of refractory depression. Since dysfunction in the frontal lobe of the brain is seen in patients with apathy, rTMS to the frontal lobe might be helpful in treating the same.

Specific Aims:

* To determine the efficacy of rTMS to the dorsolateral prefrontal cortex (DLPFC) in treating apathy in MCI in comparison to sham treatment.
* To compare the efficacy of rTMS to the DLPFC on executive function in MCI in comparison to sham treatment.

Research Plan: Current study is a randomized sham controlled cross-over study of daily rTMS.

Methods: 20 subjects with MCI and apathy will be enrolled to randomize 8 to a total of 20 sessions of treatment (2 weeks sham, 2 weeks rTMS, with 4 weeks of washout period). Subjects will be randomly assigned to rTMS or sham treatment after consent. After 2 weeks of treatment there will be a 4 week period with no treatment. At the end of the 4-week wash out period, subjects will be crossed over to the next treatment arm (i.e. those who received rTMS in the beginning will receive sham treatment and vice versa). Subjects will be followed for four additional weeks after treatment. Apathy will be assessed using the Apathy Evaluation Scale. Memory, executive function, functional status and caregiver burden will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 55 years,
2. Subjects meeting Petersen's criteria for MCI,
3. Apathy Evaluation Scale-Clinician (AES-C) score of ≥ 30,
4. Mini Mentla Status Examination (MMSE) ≥ 23,
5. Subjects who clear the TMS adult safety scale (TASS)
6. On stable dose of antidepressants (if applicable) for at least two months

Exclusion Criteria:

1. Subjects taking medications known to increase the risk of seizures from the 2012 Beers criteria: Bupropion, chlorpromazine, clozapine, maprotiline, olanzapine, thioridazine, thiothixene, and tramadol.
2. Subjects taking medications known to increase seizure threshold not listed in the Beers criteria but in the opinion of PI increase seizure threshold: tricyclic antidepressants, theophylline, methylphenidate, and high-dose thyroid supplementation.
3. Subjects taking ototoxic medications: Aminoglycosides, Cisplatin.
4. Subjects in current episode of major depression
5. History of bipolar disorder
6. Subjects with history of seizure or first degree relative with seizure disorder
7. Subjects with implanted device: wearable or implantable cardioverter defibrillators, conductive, ferromagnetic, or other magnetic sensitive metals that are implanted or are non-removable within 30 cm of the treatment coil or those with cochlear implants
8. Subjects with diagnosis of current alcohol related problems
9. Subjects with history of stroke , aneurysm, or cranial neurosurgery
10. Any condition that in the opinion of the study physician is likely to compromise their ability to safely participate in the study

Ages: 55 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (AES) | 8 weeks
  AES is an 18-item scale that assesses apathy in behavioral, cognitive and emotional domains over the previous four weeks.

SECONDARY OUTCOMES:
Trials making test | 8 weeks
  Widely used test for assessment of executive function.

OTHER OUTCOMES:
Exit 25 | 8 weeks
  EXIT-25 is a bedside measure of executive function. It defines the behavioral sequelae of executive dyscontrol and provides a standardized clinical encounter in which they can be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad R Padala, MD, MS, Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Padala PR, Padala KP, Lensing SY, Jackson AN, Hunter CR, Parkes CM, Dennis RA, Bopp MM, Caceda R, Mennemeier MS, Roberson PK, Sullivan DH. Repetitive transcranial magnetic stimulation for apathy in mild cognitive impairment: A double-blind, randomized, sham-controlled, cross-over pilot study. Psychiatry Res. 2018 Mar;261:312-318. doi: 10.1016/j.psychres.2017.12.063. Epub 2018 Jan 5. PMID 29331848